CLINICAL TRIAL: NCT00205881
Title: Bilateral Benefit in Adult Users of the HiRes 90K Bionic Ear System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AUD-BL-070705
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2012-02-10 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Hearing Loss
Keywords: HiResolution Bionic Ear; severe to profound hearing loss; bilateral implantation
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Bilaterally Implanted with HiRes 90K device.
  Interventions: Device: HiRes 90K Bionic Ear System

INTERVENTIONS:
Device: HiRes 90K Bionic Ear System — Cochlear implant system

SUMMARY:
Normal hearing listeners gain important everyday benefits from listening with two ears (bilateral hearing) compared to their baseline performance with hearing aids. Advantages of bilateral hearing include the ability to determine where sounds are coming from and the ability to hear sounds and understand speech in noisy environments. Based upon these advantages, this study will (1) evaluate the benefit of hearing with two Bionic Ear implants (one in each ear) and (2) compare HiResolution sound processing with conventional sound processing.

ELIGIBILITY:
Inclusion Criteria:

1. No previous implant experience.
2. Age 18 years or older.
3. Postlingual onset of hearing loss.
4. Sensorineural hearing loss of a severe or greater degree in both ears.
5. Normal/patent cochlear anatomy in each ear.
6. English language proficiency.
7. Willingness and ability to participate in all scheduled procedures.

Exclusion Criteria:

No exclusion criteria specified, except for the opposite of inclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Joe Osberger, Study Chair — Advanced Bionics
Locations (9):
- United States (9):
  - House Clinic/House Ear Institute, Los Angeles, California
  - California Ear Institute (Let Them Hear Foundation), Palo Alto, California
  - University of Miami - Cochlear Implant Center, Miami, Florida
  - Tampa Bay Hearing and Balance Center, Tampa, Florida
  - Carle Clinic Association, Urbana, Illinois
  - Spectrum Health, Grand Rapids, Michigan
  - Midwest Ear Institute, Kansas City, Missouri
  - New York University Cochlear Implant Center, New York, New York
  - Dallas Otolaryngology Associates, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Bilaterally Implanted: 31 Subjects were bilaterally implanted with Bionic ear systems within the same surgery. 1 Subject was unilaterally implanted.
Period: Overall Study
Arm/Group | Bilaterally Implanted
Started | 32
Completed | 16 (32 enrolled. 1 unilateral. 25 bilateral for data analysis at 8 months. 16 completed study.)
Not Completed | 16
Not completed — Withdrawal by Subject | 16

BASELINE CHARACTERISTICS:
Arm/Group | Bilaterally Implanted
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 52.6 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Pre-implant Consonant-Nucleus-Consonant (CNC) Scores to Post-implant CNC Scores in Bilateral Users.
Description: Participants were tested on 50 monosyllabic, phonetically balanced words from the Consonant-Nucleus-Consonant (CNC) set, prior to implantation and after bilateral implantation. Percent correct scores for the CNC test are reported.
Time Frame: 8 months of bilateral cochlear implant use
Population: Adults with severe-to-profound hearing loss who received bilateral cochlear implants in the same operation.
Measure: Mean (Standard Deviation); unit: percent of words correct
Groups:
- Baseline: Testing with hearing aids in best-aided condition.
- 8 Months Post-device Activation: Testing conducted with bilateral implants.
Arm/Group | Baseline | 8 Months Post-device Activation
Number analyzed (Participants) | 24 | 25
percent of words correct | 4.0 (8.0) | 69.0 (23.0)

2. Secondary Outcome: HINT Sentences in Noise
Description: 20 sentences presented in noise at fixed levels
Time Frame: 8 months of bilateral cochlear implant use
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Bilaterally Implanted
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 7/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilaterally Implanted (N=31)
Dizziness (Ear and labyrinth disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators were not permitted to disclose study results until the Sponsor had completed data analyses and report generation for regulatory purposes, and/or received regulatory approval. The Sponsor agreed to notify the Investigators when they were free to publish, present or use any results arising out of this study for their own instructional, research, or publication objectives, provided that such publication did not disclose any of the Sponsor's proprietary information.